CLINICAL TRIAL: NCT05737888
Title: Physiological Regulation of Chronic Tinnitus
Acronym: NeuroTin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyss Center for Bio and Neuroengineering (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeuroTin
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Tinnitus
Keywords: Tinnitus; EEG neurofeedback; fMRI neurofeedback; Cognitive behavioral therapy
MeSH Terms: conditions — Tinnitus | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Prospective research with 3 independent research arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fMRI Neurofeedback (Experimental): The participants receive visual feedback (displayed on a screen) related to BOLD activity from their auditory cortices, and they are asked to learn to down-regulate it.
  Interventions: Other: fMRI Neurofeedback
- EEG Neurofeedback (Experimental): The participants receive visual feedback (displayed on a screen) related to the ratio of alpha to delta localized activity from their auditory cortices, and they are asked to learn to up-regulate it.
  Interventions: Other: EEG Neurofeedback
- Cognitive Behavioral Therapy (Active Comparator): Group therapy is provided by trained clinicians for research participants. Participants are confronted with tinnitus-inducting situations and trained to use diverse cognitive and behavioral coping skills to reduce the subjective impact of tinnitus burden. Such coping skills include relaxation, distraction, and de-catastrophizing, among other strategies.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Other: fMRI Neurofeedback — 15 intervention sessions on a 3T MRI scanner.
  Arms: fMRI Neurofeedback
Other: EEG Neurofeedback — 15 intervention sessions with a standard EEG-cap with 64 active electrodes.
  Arms: EEG Neurofeedback
Behavioral: Cognitive Behavioral Therapy — 10 intervention sessions of CBT group therapy, as per local university hospital standard of care.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The present project involves research on humans with the aim to characterize the reduction of chronic, continuous, non-pulsatile and debilitating tinnitus in humans by comparing neurofeedback (fMRI or EEG) to the current gold standard behavioral cognitive therapy.

DETAILED DESCRIPTION:
Chronic tinnitus is affecting 10-15% of people typically for many decades, with increasing prevalence with aging. Multiple therapy forms for tinnitus exist (including cognitive behavioral therapy, external white noise stimulation, meditation, and various kinds of alternative approaches), but up to now, no generally accepted successful treatment exists. Previously, it was shown that voluntary control of the activation of the auditory cortex can be learned by means of real-time functional Magnetic Resonance Imaging (fMRI) neurofeedback, and that it may alleviate tinnitus symptoms. The same seems to hold for learned increase of alpha activity localized in the auditory cortex through electroencephalography (EEG) neurofeedback. Given the high prevalence of chronic tinnitus, its significant burden for affected individuals, and given the absence of generally effective therapy, neurofeedback training for tinnitus has the potential to become a clinical application.

The main goal of this project is to comparatively assess tinnitus reduction using neurofeedback (fMRI or EEG) compared to cognitive behavioral therapy in participants with chronic severe tinnitus.

* The participants are assigned to 3 different experimental groups (EEG neurofeedback, fMRI neurofeedback, or cognitive behavioral therapy). The participation per subject will last from 4 to 12 months.
* The participants undergo medical tests including audiological tests as well as questionnaires related to tinnitus and quality of life at different timepoints of the study (pre and post training visits).
* At the end of the experimental visits, each participant will have one early and one late post-assessment evaluation visits.
* In order to evaluate the longer-term evolution of tinnitus over time, long-term follow-ups will be scheduled starting at 9 months after the final experimental visit, and will occur every 4.5 months thereafter, until research ends (for a maximum of 5 years).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 80 years
2. Tinnitus Handicap Inventory ≥ 48
3. Chronic, persistent, non-pulsatile tinnitus for minimum 6 months
4. Functional hearing
5. Normal inner ear structure assessment using an ear microscope, normal tympanic membrane mobility
6. Participant willing, able and available to participate in the entire research, including completion of questionnaires and traveling to research sites for the duration of the trial

Exclusion Criteria:

1. Contraindication to MRI (e.g. non compatible cochlear implant, pacemaker, deep brain stimulation)
2. Conductive hearing loss exceeding 20 dB at two or more frequencies
3. Known diagnoses causing tinnitus or hearing loss:

   * Known systemic disease (vestibular schwannoma, endolymphatic hydrops)
   * Lesion in central nervous system, including history of severe cranio-cerebral trauma
   * Acute ear canal or middle ear inflammation or effusion
4. Significant neurologic disease, psychiatric disease, substance abuse or acute allergic disease
5. Ongoing medication that is known to treat, influence, or cause tinnitus (e.g. high-dose aspirin, quinidine, aminoglycosides)
6. Ongoing or recent (completed since less than 4 weeks) tinnitus therapy (e.g. tinnitus maskers, acupuncture)
7. Participation in competitive or pharmacological study
8. Pregnant woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Behavioral improvement of tinnitus as measured by the Tinnitus Handicap Inventory (THI) | 8 months
  To show that behavioral improvement of tinnitus after intensive neurofeedback training is equivalent or better than improvement obtained after attending group cognitive behavioral therapy, as measured by Tinnitus Handicap Inventory (THI) scores reported before experiment and at late post-assessment (significant difference, p-value < 0.05). THI ranges from low scores (grade 1 - slight or no handicap), to highest scores (grade 5 - catastrophic handicap).

SECONDARY OUTCOMES:
Audiological measures | 8 months
  If reported tinnitus scores correlate with audiological measures during research for each experimental group;
Training effect | 8 months
  If significant behavioral change as shown by a THI grade reduction is observed before/after experiment in each group;
Other factors | 8 months
  If there are external parameters influencing reported tinnitus levels for each group during the research, based on participant questionnaires (i.e., placebo effect of the trainer/CBT professional provider, motivation levels);
Correlation with BOLD signal | 8 months
  Specifically for group 1 - fMRI neurofeedback, whether evolution of audiological and tinnitus measures at different research timepoints correlate with BOLD signal of the auditory cortex;
Correlation with alpha activity | 8 months
  Specifically for group 2 - EEG neurofeedback, whether evolution of audiological and tinnitus measures at different research timepoints correlate with alpha activity of the auditory cortex;
Acceptance of intensive schedule | 8 months
  Specifically for group 1 and 2, acceptance of neurofeedback intensive schedule of visits by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Senn, MD, PhD, Principal Investigator — Dept. of Otology, Audiology and Cochlear Implant Surgery, University Hospital Geneva
Locations (1):
- Dept. of Otology, Audiology and Cochlear Implant Surgery, University Hospital Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gninenko N, Trznadel S, Daskalou D, Gramatica L, Vanoy J, Voruz F, Robyn CL, Spadazzi A, Yulzari A, Sitaram R, Van De Ville D, Senn P, Haller S. Functional MRI Neurofeedback Outperforms Cognitive Behavioral Therapy for Reducing Tinnitus Distress: A Prospective Randomized Clinical Trial. Radiology. 2024 Feb;310(2):e231143. doi: 10.1148/radiol.231143. PMID 38349241